CLINICAL TRIAL: NCT02569554
Title: A Phase 1, Randomized, Crossover, Open-Label, 4 Period Study In Healthy Volunteers To Demonstrate The Lack Of Effect Of Rabeprazole And Food On The Pharmacokinetics Of PF-06463922 And To Assess The Relative Bioavailability Of Oral Solution To The Tablet Formulation Of PF-06463922
Brief Title: PPI And Food Effect Study For PF-06463922 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7461008; 2015-003416-21 (EudraCT Number); PPI STUDY (Other: Alias Study Number)
Record Dates: First submitted 2015-10-05; First posted 2015-10-06 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: PF-06463922; rabeprazole; proton pump inhibitor (PPI); pharmacokinetics(PK); food effect
MeSH Terms: interventions — lorlatinib; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-06463922 (Experimental): each subject will receive four single doses of PF-06463922 without food, with food, with rabeprazole (without food), and one of the two new formulations without food.
  Interventions: Drug: PF-06463922; Drug: rabeprazole

INTERVENTIONS:
Drug: PF-06463922 — each subject will receive 4 single oral doses of 100 mg PF-06463922 (treatment A: tablets without food; treatment B: tablets with food; treatment C: tablets without food with rabeprazole; treatment D: oral solution without food). There will be at least 10 days washout period between consecutive PF-06463922 single dose.
Drug: rabeprazole — 20 mg daily tablets in the evening for 5 days and Pf-06463922 on the morning of day 6 in treatment C.
  Other Names: Pariet

SUMMARY:
The current study will be conducted in healthy adult subjects to evaluate the effect of proton pump inhibitor and food on pharmacokinetics of PF-06463922, to evaluate the bioavailability of the oral solution relative to the tablet formulation of PF-06463922.

DETAILED DESCRIPTION:
PF-06463922 is a selective, ATP competitive small molecule tyrosine kinase inhibitor (TKI) of the Anaplastic Lymphoma Kinase (ALK) positive (ALK+) or ROS oncogene 1 (ROS1) positive (ROS1+) receptor tyrosine kinases (RTK) that also potently inhibits ALK kinase domain mutations responsible for resistance to crizotinib. PF-06463922 is being developed as a novel anticancer agent for the treatment of patients with advanced ALK+ NSCLC or ROS1+ NSCLC.

The current study is a Phase 1, randomized, open label, 4 period, 4 treatment, 4 sequence, crossover study conducted in healthy adult subjects. Each subject will receive four single oral doses of 100 mg PF-06463922 as tablets alone, tablets with food, tablets with rabeprazole, and oral solution after overnight fasting with at least a 10 day washout period between each PF-06463922 dose.

Twenty four (24) subjects will be enrolled to obtain at least 20 evaluable subjects who complete all treatments. Subjects who withdraw will not be replaced unless the total number of completed subjects falls below 20.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non-childbearing potential and/or male subjects
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document.
* Subject must be willing to avoid direct sunlight exposure or any high intensity ultraviolet light exposure

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular
* Any condition possibly affecting drug absorption
* A positive urine drug screen.
* Use of tobacco- or nicotine containing products within 90 days of screening or a positive urine cotinine test and history of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males within 6 months of Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
plasma AUCinf for PF-06463922 | 3 months
  area under plasma concentration-time profile from time 0 extrapolated to infinite time for PF-06463922
plasma Cmax for PF-06463922 | 3 months
  observed maximal plasma PF-06463922 concentration

SECONDARY OUTCOMES:
plasma AUClast for PF-06463922 | 3 months
  area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration for PF-06463922
plasma Tmax for PF-06463922 | 3 months
  time to the plasma maximal concentration for PF-06463922
plasma t1/2 for PF-06463922 | 3 months
  plasma terminal half-life for PF-06463922
plasma CL/F for PF-06463922 | 3 months
  apparent clearance for PF-06463922
plasma Vz/F for PF-06463922 | 3 months
  apparent volume of distribution for PF-06463922

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7461008&StudyName=A%20Phase%201%2C%20Randomized%2C%20Crossover%2C%20Open-label%2C%204%20Period%20Study%20In%20Healthy%20Volunteers%20To%20Demonstrate%20The%20Lack%20Of%20Effect%20Of%20Rabeprazole%20And%20Food%20On%20The%20Pharmacokinetics%20Of%20Pf-06463922%20And%20To%20Assess%20The%20Relative%20Bioavailability%20Of%20Oral%20Solution%20To%20The%20Tablet%20Formulation%20Of%20Pf-06463922